CLINICAL TRIAL: NCT01292499
Title: Italian Network for the Improvement of Compliance in Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ospedale Amedeo di Savoia (Other)
Responsible Party: Carmine Munizza, Centro Studi e Ricerche in Psichiatria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RIMAT-De; RIMAT-De
Record Dates: First submitted 2011-01-26; First posted 2011-02-09 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2010-12

CONDITIONS: Depression
Keywords: psychotherapy; psychoeducation; depression
MeSH Terms: conditions — Depression | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Pharmacological treatment (No Intervention): Pharmacological treatment consists of the administration of a single antidepressant drug. The treatment will be administered as currently done by the mental health center, taking into due account patient's age, general health, previous response to antidepressant drugs, comorbidity, and potential side effects of drugs.
- Psychotherapy (Experimental): Will receive psychotherapy as well (10 sessions). Psychoterapy will consist of 10 weekly sessions, lasting about 50 minutes each. Psychotherapy will begin after 4-6 weeks from the beginning of the pharmacological treatment, to allow drugs to be effective. The overall list of visits scheduled for the patients is defined during the second psychiatric visit, to allow a reasonable planning of all of the appointments required for that particular patient. Psychotherapists will be free to follow the approach they were trained.
  Interventions: Behavioral: Psychotherapy
- Psychoeducation (Experimental): Will receive psychoeducation as well, with phone monitoring and regular follow-ups. Psychoeducation does not simply mean making the patient aware of depression etiology and drugs effect. In fact, patients should receive additional counselling about how to integrate the pharmacological treatment in their daily routine and to solve possible problems, in order to allow them to be actively and constantly involved in the treatment they are going to receive. Patients will receive 7 sessions of psychoeducation and 7 phone calls during the first 5 months. In addition, all of the patients will receive a brochure explaining the most important aspects of their disorder.
  Interventions: Behavioral: Psychoeducation
- Psychoeducation and psychotherapy (Experimental): Will receive both psychoeducation and psychotherapy sessions.
  Interventions: Behavioral: Psychoeducation and psychotherapy

INTERVENTIONS:
Behavioral: Psychotherapy — 10 sessions (50 min)
  Arms: Psychotherapy
Behavioral: Psychoeducation — 7 sessions + 7 phone calls
  Arms: Psychoeducation
Behavioral: Psychoeducation and psychotherapy — Psychoeducation + psychotherapy
  Arms: Psychoeducation and psychotherapy

SUMMARY:
The RIMAT-De study (Rete Italiana per il Miglioramento dell'Adesione al Trattamento nella Depressione) is a multicentric Randomized Controlled Clinical Trial aiming at identifying the best strategies available to reduce the poor compliance of patients with antidepressant drugs. Patients' compliance will be measured within six months of pharmacological treatment, comparing the specific contributions of brief psychotherapy and psychoeducational interventions: the psychoeducational intervention will encompass the monitoring of drugs' side effects and patients' satisfaction. In the rest of the document, for the sake of brevity the two treatments previously described will be indicated as "psychotherapy" and "psychoeducation". These treatments will be compared with the treatment usually carried on by the mental health centers involved (i.e. treatment as usual, TAU). The factorial design of the study will take into consideration the combination of the two treatments (i.e. psychotherapy and psychoeducation) as well.

DETAILED DESCRIPTION:
Another important aim of the study is the investigation of whether the clinical improvement depends on the efficacy of the psychological treatments proposed per se, or whether they just contribute to increase the compliance with the pharmacological treatment, maintaining the patients on treatment longer and allowing the drugs to reach long-lasting effects. While recognizing the general therapeutic efficacy of psychotherapy in the treatment of depressive disorders, nevertheless the present study aims at verifying whether an equal therapeutic effect may be reached via a better compliance with the pharmacological treatment, fostered for example by the psychoeducational intervention. The rationale lays on the ease of transferability of psychoeducational interventions to the general clinical practice, that usually suffers from lack of resources in implementing structured psychotherapy interventions.

ELIGIBILITY:
Inclusion Criteria:

1. New episode of depression, according to the DSM-IV (Codes F32 Major Depressive Disorder, single episode; F33 Major Depressive Disorder, recurrent; F34.1 Dysthymic Disorder; F32.9 Depressive Disorder, not otherwise specified), or new contact with the Mental Health Center for recurrent depression (same Codes) after a six-month period (or longer) without any treatment;
2. Age >= 18 years old;
3. QIDS-SR16 score >=10;
4. Necessity of a pharmacological antidepressant treatment;
5. Written informed content given by the participant before the beginning of the study.

Exclusion Criteria:

1. Comorbidity of schizophrenic disorder, according to the DSM-IV (Codes F06.3 - Organic mood disorder; F20 - Schizophrenia; F29 -Uunspecified Nonorganic Psychosis; F30-F31 - Manic Episode and Bipolar Affective Disorder; F34.0 - Cyclothymia; F10-F19 - Mental and Behavioural Disorders due to Psychoactive Substance Use).
2. Current pregnancy.
3. Probable hospitalization, for whatever reason.
4. Patient seen once and then referred to his/her GP or other specialist physician;
5. Pharmacological treatment already prescribed by a psychiatry or neurology specialist. However, if the patient is not satisfied with the current treatment and/or the psychiatrist involved in the present study considers appropriate to change the treatment, the present exclusion criterion will not be valid any longer.
6. Pharmacological treatment prescribed for more than 15 days by patient's GP. However, if the patient is not satisfied by the treatment and/or the psychiatrist involved in the present study considers appropriate to change the treatment, the present exclusion criterion will not be valid any longer.
7. The patient is currently under psychotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1264 (Estimated)
Dates: Start 2009-03; Primary Completion 2012-01 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients showing good compliance, as measured at six months from the beginning of the treatment. | 3 years
  The effect size is conceptualized as the difference between the proportion of patients in the 4 treatment arms showing good compliance at the end of the study. The effects of the two treatments (psychotherapy and psychoeducation) will be measured separately, via stratified analyses and multivariate regression models, as appropriate.

CONTACTS AND LOCATIONS:
Locations (1):
- ASL TO2 Amedeo di Savoia, Torino, Torino, Italy